CLINICAL TRIAL: NCT03516305
Title: A Phase 1 Open-Label, Non-Randomized, Single-Dose, Pharmacokinetic Study Evaluating Staccato® Alprazolam 1 mg Inhaler in Smoker Versus Non-Smoker Healthy Adult Volunteers
Brief Title: Pharmacokinetic Study Evaluating Staccato® Alprazolam 1 mg Inhaler in Smokers Versus Non-Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Engage Therapeutics, Inc. (Industry)
Collaborators: Clinilabs, Inc. (Other)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EPK-002
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: All subjects receive a single dose of Staccato Alprazolam 1 mg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Staccato Alprazolam 1 mg (Experimental): a single inhaled dose
  Interventions: Drug: Staccato Alprazolam 1 mg

INTERVENTIONS:
Drug: Staccato Alprazolam 1 mg — alprazolam I mg administered via the Staccato hand-held inhaler device system.

SUMMARY:
This is an open-label, non-randomized, single dose, pharmacokinetic study in 36 healthy adult male and female volunteers, including 18 smokers and 18 non-smokers. All subjects will be administered a single inhaled dose of Staccato alprazolam 1 mg via hand-held inhaler. Blood samples will be drawn for pharmacokinetic analysis. Eligible subjects are admitted to Phase 1 unit for up to 48 hours. Subjects will receive a post-study safety phone call 14 days(± 2 days) after dosing.

ELIGIBILITY:
Inclusion Criteria:

* These inclusion criteria (items 1-8) apply to all subjects, smokers and non-smokers:

I. Healthy male and female subjects between the ages of21 to 50 years, inclusive.

2. Body mass index (BMI) >/= 18 and </= 30 kg/m2, inclusive.

3. Able to speak, read, and understand English and are willing and able to provide written informed consent on an IRB-approved form prior to the initiation of any study procedures.

4. Willing and able to be confined to a clinical research facility for up to 48 hours (including 2 nights) and comply with the study schedule and study requirements.

5. Normal spirometry at screening as demonstrated by FEVI +/- 80% of predicted and FVC +/- 80% of predicted.

6. Adequate veins, as assessed by the Investigator or Investigator's designee, that are suitable for the required number and frequency of PK blood draws in this study.

7. In otherwise good general health as determined by a complete medical history, physical examination, 12-lead electrocardiogram (ECG), blood chemistry profile, hematology, serology (HIV-l/2Ab, HBsAg, HCV Ab), and urinalysis at screening.

8. Female participants (if of child-bearing potential and sexually active) and male participants (if sexually active with a partner of child-bearing potential) who agree to use a medically acceptable and effective birth control method throughout the study and for one week following the end of the study.

Smokers must meet the following inclusion criteria (items 9-10):

9. A history of smoking> 15 cigarettes/day currently and for at least the last 2 years.

10. Serum cotinine +/-500 ng/mL at Screening Visit I.

Nonsmokers must meet the following inclusion criteria (items 11-12):

11. A history of never smoking> 5 cigarettes/day and not smoking at all for at least the last 2 years prior to Visit I.

12. Serum cotinine :o 40 ng/mL at Screening Visit I and a negative urine cotinine test at Visit 2 Day-I.

Exclusion Criteria:

1. Treatment with an investigational drug within 30 days ( or within 5 half-lives of the investigational drug, if>30 days) prior to Visit I.
2. Significant hepatic, renal, gastroenterologic, cardiovascular endocrine, neurologic (including history of seizures or stroke), or hematologic disease.
3. Any acute illness in the 5 days prior to Visit 2.
4. Upper respiratory tract infection within 6 weeks of Visit 2 or bronchitis or pneumonia within 6 months of Visit 2.
5. Use of a bronchodilator for the treatment of wheezing within 12 months of Visit I.
6. Diagnosis of an active or chronic pulmonary disease.
7. Lung resection or other pulmonary surgery within 12 months of Visit I.
8. A history of allergy or intolerance to alprazolam.
9. Use of any other prescription or nonprescription medication--with the exception of acetaminophen, ibuprofen or ongoing doses of oral contraceptives or vitamins--within 5 days prior to study drug administration.
10. A history within the past 2 years of drug or alcohol dependence or abuse.
11. Positive test for alcohol or a positive urine screen for drugs of abuse at screening
12. A positive HIV test.
13. Breastfeeding or a positive pregnancy test at screening (female subjects).
14. Clinically significant ECG abnormality.
15. Hypotension or hypertension, at screening or baseline.
16. Poor veins in the opinion of the Investigator or the Investigator's designee such that the participant is judged to likely have difficult venipuncture during the study.
17. Any other disease or condition, by history, physical examination, or laboratory abnormalities that in the investigator's opinion, would present undue risk to the subject, or may confound the interpretation of study results.
18. Participation in another clinical trial within 2 months of the beginning of the present study, or blood donation or comparable blood loss (>350mL) within 2 months before the present study.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) : Maximum observer drug concentration (Cmax) | Sequential time points : pre-dose, and at 2, 5, 10 and 30 minutes, and at 1, 2, 4, 6, 12, 24 and 36 hours post-dose.
  Cmax of alprazolam in smokers compared to non-smokers
PK: Area under the concentration versus time curve (AUC)from Zero to Infinity (AUC[0-∞] | Sequential time points : pre-dose, and at 2, 5, 10 and 30 minutes, and at 1, 2, 4, 6, 12, 24 and 36 hours post-dose.
  AUC[0-∞] of alprazolam in smokers compared to non-smokers

SECONDARY OUTCOMES:
PK;: time after administration of a drug when the maximum plasma concentration is reached (Tmax) | Sequential time points : pre-dose, and at 2, 5, 10 and 30 minutes, and at 1, 2, 4, 6, 12, 24 and 36 hours post-dose.
  Tmax of alprazolam in smokers compared to non-smokers
PK: half-life (t1/2) | Sequential time points : pre-dose, and at 2, 5, 10 and 30 minutes, and at 1, 2, 4, 6, 12, 24 and 36 hours post-dose.
  t1/2 of alprazolam in smokers compared to non-smokers

CONTACTS AND LOCATIONS:
Overall Officials: M. Shenouda, MD, Principal Investigator — Clinilabs, Inc.
Locations (1):
- Clinilabs Research Unit, Eatontown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No